CLINICAL TRIAL: NCT01353443
Title: Prophylactic Mesh Implantation After Abdominal Aortic Aneurysm Repair. A Prospective, Randomised, Controlled Study
Brief Title: Prophylactic Mesh Implantation After Abdominal Aortic Aneurysm Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: AIDA Study
Record Dates: First submitted 2011-04-18; First posted 2011-05-13 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm; AAA
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (No Intervention): Monofilament absorbable MonoPlus® suture material will be used for closing of the midline incision.
- Group B (Other): Abdominal wall closure with monofilament absorbable MonoPlus® suture material and onlay placement of Optilene® Mesh Elastic fixed by sutures.
  Interventions: Procedure: Optilene® Mesh Elastic
- Group C (No Intervention): Monofilament, absorbable MonoMax suture material will be used for the closure of the abdominal cavity.

INTERVENTIONS:
Procedure: Optilene® Mesh Elastic — A number of patients will receive a Optilene® Mesh Elastic mesh, which may not be clinically indicated.
  Arms: Group B

SUMMARY:
AIDA Study is a prospective, multicentre, randomized, controlled clinical investigation with patients undergoing median laparotomy for Abdominal Aortic Aneurysm (AAA) repair.

The primary objective of the clinical investigation is to test the hypothesis that insertion of an Optilene® Mesh Elastic mesh - a monofilament, light-weight, large pore sized, polypropylene mesh manufactured by Aesculap AG - is superior to suturing alone and will reduce the hernia formation rate within the first 2 years.

A reduction from 30% to 10% of the patient population is assumed.

DETAILED DESCRIPTION:
One of the late complications of the elective surgery of an Abdominal Aortic Aneurysms (AAA) is the formation of an incisional hernia following the AAA repair.

The high frequency of incisional hernia formation in the AAA patients suggests the presence of a structural defect within the fascia.

As a result of these information and that obtained from a small pilot study using mesh prophylactically in high risk group of patients, the concept of using a mesh prophylactically for AAA repairs seems an area worth further exploration.

Owing to the availability of the new generation of meshes with proven good biocompatibility it would seem that this could be a viable means of reducing the herniation rate and therefore re-operation in this high risk population.

Within the investigation Patients requiring elective surgical repair of an AAA will be randomized in one of the following three different groups:

* Group A: Monofilament absorbable MonoPlus® suture material will be used for closing of the midline incision.
* Group B: Abdominal wall closure with monofilament absorbable MonoPlus® suture material and onlay placement of Optilene® Mesh Elastic fixed by sutures.
* Group C: Monofilament, absorbable MonoMax® suture material will be used for the closure of the abdominal cavity.

A total of 282 patients who meet the eligibility criteria will be entered into the clinical investigation (Group A = 94 patients, Group B = 94 patients and Group C = 94 patients).

All patients will have follow-up clinical visits 2 days after surgery, at day of discharge, at 3, 6, and 12 months and a final visit at 24 months. All patients will be asked to complete the health status patient questionnaire EQ-5D preoperatively and at 3, 6, 12 and 24 months postoperatively. As all patients routinely receive an ultrasound at 3, 6, 12, and 24 months, this information will be used to confirm if a hernia is present.

The primary objective of the clinical investigation is to test the hypothesis that insertion of an Optilene® Mesh Elastic mesh is superior to suturing alone and will reduce the hernia formation rate within the first 2 years.

Secondary objectives include:

1. Lower herniation rate in the 12 months after mesh implantation in group B as compared to group A
2. Non-inferiority of MonoMax suture material (group C) in comparison to MonoPlus suture material (group A) concerning the rate of incisional hernia after abdominal wall closure at 3, 6, 12, and 24 months after surgery.
3. Mean time, in days, to return to normal activities as determined by CRF question (comparison of groups A, B, C).
4. Mean time, in days, to return to work as determined by CRF question (comparison of groups A, B, C).
5. Differences in mean patient health status as determined by using a patient questionnaire (EQ-5D) at 3, 6, 12 and 24 months post-operatively; pre-operative baseline will be recorded (groups A-C).
6. Number of wound complications (groups A-C) as determined by medical assessment post-operatively immediately prior to discharge, and at the clinical visits at 3, 6, 12 and 24 months, including infections, seromas, haematomas, and hernia formation, confirmed by ultrasound examination.
7. Safety as determined by collection of adverse events in the CRF (groups A-C).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients >18 years of age.
2. Patients undergoing an elective surgery for AAA repair.
3. Patients who currently have no malignant disease requiring therapy.
4. Patients who are able to fulfill all clinical investigation requirements
5. Patients who have provided written informed consent.

Exclusion Criteria:

1. Patients who require median laparotomy for AAA repair as an emergency procedure.
2. Expected length of fascia incision > 30 cm.
3. Patients with coagulopathy
4. Patients who have had previous median laparotomy and/or laparotomy crossing the incision necessary for AAA laparotomy.
5. Patients with current immunosuppressive therapy (>40 mg corticoid/day or azathioprine).
6. Chemotherapy within the last 4 weeks.
7. Radiotherapy on the treated region within the last 2 months.
8. Pregnant and breast-feeding women.
9. Known allergy against ingredients of the investigational products (polypropylene, poly-4-hydroxybutyrate, polydioxanone).
10. Patients participating in other investigational drug or medical device studies within the preceding 4 weeks.
11. Patients with an ongoing medical condition or social reason that may affect their ability to complete the two years follow-up period.
12. Life expectancy less than 24 months.
13. Severe psychiatric or neurologic disease.
14. Lack of compliance.
15. Drug abuse.
16. Inability to understand and follow the instructions given by the investigator (e.g. dementia, lack of time, insufficient command of language).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2011-02; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Herniation rate | 24 months
  As an indicator of efficacy, the reduction of herniation rate will be verified by clinical examination and confirmed by Ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Debus, Prof. Dr., Principal Investigator — University Heart Center Hamburg - Eppendorf
Locations (9):
- Germany (9):
  - Klinikum Stuttgart - Katharinenhospital (KH), Stuttgart, Baden-Wurttemberg
  - Klinikum Nürnberg Süd, Nuremberg, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia
  - Klinikum Bremen-Nord, Bremen
  - University Heart Center Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Wandsbek, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Klinikum Ludwigsburg, Ludwigsburg

REFERENCES:
- [Result] Honig S, Diener H, Kolbel T, Reinpold W, Zapf A, Bibiza-Freiwald E, Debus ES; for AIDA study group. Abdominal incision defect following AAA-surgery (AIDA): 2-year results of prophylactic onlay-mesh augmentation in a multicentre, double-blind, randomised controlled trial. Updates Surg. 2022 Jun;74(3):1105-1116. doi: 10.1007/s13304-021-01125-0. Epub 2021 Jul 21. PMID 34287760